CLINICAL TRIAL: NCT02230436
Title: The Impact of Early Versus Late Drain Removal on Postoperative Morbidity After Pancreatectomy: A Randomized Prospective Trial
Brief Title: Early Versus Late Drain Removal After Pancreatectomy: A Randomized Prospective Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-GS02
Record Dates: First submitted 2014-08-16; First posted 2014-09-03 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-08

CONDITIONS: Pancreatectomy; Post Procedural Discharge
Keywords: Pancreatectomy; Time of drain removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early drain removal (Experimental): Removing drain(s) on postoperative day 3 (n = 72)
  Interventions: Other: Early drain removal
- Late drain removal (Experimental): Removing drain(s) on postoperative day 4 or later (n = 72)
  Interventions: Other: Late drain removal

INTERVENTIONS:
Other: Early drain removal — Removing drain(s) on postoperative day 3
  Arms: Early drain removal
Other: Late drain removal — Removing drain(s) on postoperative day 4 or later
  Arms: Late drain removal

SUMMARY:
The aim of this study is to demonstrate the hypothesis that early removal of drain can reduce the incidence of intra-abdominal infection and pancreatic fistula after pancreatectomy compared with later removal of drain.

DETAILED DESCRIPTION:
This study is to analyze the association between the time of removal of drain after pancreatic resection and incidence of intra-abdominal complications, such as intra-abdominal infection and pancreatic leakage. We design a prospective randomized study. Patients with pancreatic and periampullar tumors who underwent pancreatoduodenectomy (PD) or distal pancreatectomy (DP) are recruited to the study if amylase value in drain(s) is less than 5000 U/L on postoperative day (POD) 1. After obtaining informed consent, eligible patients are randomly allocated to early or late drain removal group on POD 3. In the group A, drain(s) are removed on POD 3, whereas in group B drain is removed on POD 4 or beyond. The primary outcomes are the incidence of intra-abdominal infection and pancreatic fistula; the secondary outcomes include intra-abdominal bleeding, delayed gastric emptying, pulmonary complications, and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age: >18yr, <75yr
* Patients with pancreatic diseases (including tumor and inflammatory disease) or non-pancreatic tumors (biliary duct cancer or ampullary tumor) who underwent pancreatoduodenectomy (PD) or distal pancreatectomy (DP)
* The amylase value in drain(s) is less than 5000 U/L on postoperative day 1 and 3.

Exclusion Criteria:

* Reconstruction of the pancreatic remnant by pancreaticogastrostomy
* Intra-abdominal hemorrhage within 72 hours after operation
* Biliary fistula (output of biliary fluid from at least 1 abdominal drain) within 72 hours after operation
* Chylous leakage (milky water) within 72 hours after operation
* The volume of drain effluent (ascites) is greater than 300 ml within 72 hours after operation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Intra-abdominal infection | Up to postoperative 30 days
  Positive cultures of collection of fluid or blood,or persistent fever necessitating treatment with antibiotics and positive detection in image test.
Pancreatic fistula | Up to postoperative 30 days
  The international study group (ISGPF) definition: A drain output of any measurable volume of fluid on or after postoperative day 3 with an amylase content greater than 3 times the serum amylase activity. Three different grades of postoperative fistula (grades A, B, C) are defined according to the clinical impact on the patient's hospital course.

SECONDARY OUTCOMES:
Intra-abdominal bleeding | Up to postoperative 30 days
  The International Study Group of Pancreatic Surgery (ISGPS) definition: Blood loss through abdominal drains or nasogastric tube;hematemesis or melena; clinical deterioration of the patient; unexplained hypotension or tachycardia; or laboratory findings such as a decreasing hemoglobin concentration.
Delayed gastric emptying | Up to postoperative 30 days
  The International Study Group of Pancreatic Surgery (ISGPS) definition: Inability to return to a standard diet by the end of the first postoperative week with prolonged nasogastric intubation.
Pulmonary complications | Up to postoperative 30 days
  Including pulmonary infection and atelectasis.
Length of hospital stay (day) | Up to postoperative 2 weeks
  Participants will be followed for the duration of hospital stay, an expected average of 2 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Menghua Dai, M.D., Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Background] Wente MN, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Traverso LW, Yeo CJ, Buchler MW. Delayed gastric emptying (DGE) after pancreatic surgery: a suggested definition by the International Study Group of Pancreatic Surgery (ISGPS). Surgery. 2007 Nov;142(5):761-8. doi: 10.1016/j.surg.2007.05.005. PMID 17981197
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Background] Wente MN, Veit JA, Bassi C, Dervenis C, Fingerhut A, Gouma DJ, Izbicki JR, Neoptolemos JP, Padbury RT, Sarr MG, Yeo CJ, Buchler MW. Postpancreatectomy hemorrhage (PPH): an International Study Group of Pancreatic Surgery (ISGPS) definition. Surgery. 2007 Jul;142(1):20-5. doi: 10.1016/j.surg.2007.02.001. PMID 17629996